CLINICAL TRIAL: NCT01914900
Title: Phase II Study of Preoperative TPF Chemotherapy in Locally Advanced Resectable Oral Cavity Squamous Cell Cancer in Order to Improve the Rate of Pathological Complete Response
Brief Title: Preoperative TPF Chemotherapy in Molecularly Selected Locally Advanced Resectable Oral Cavity Squamous Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Lisa Licitra, MD, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT40/10
Record Dates: First submitted 2013-07-29; First posted 2013-08-02 (Estimated); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Locally Advanced Resectable Oral Cavity Squamous Cell Cancer
Keywords: oral cavity cancer; induction chemotherapy; TP53; beta tubulin II
MeSH Terms: conditions — Mouth Neoplasms | interventions — Docetaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- induction TPF chemotherapy (Experimental): Each patient will receive induction CT, consisting of TPF (docetaxel 75 mg/sm and cisplatin 80 mg/sm day 1 and 5 fluorouracil 800 mg/sm each day in continuous infusion day 1-4, according to Paccagnella et al, ASCO 2008) for 3 cycles every 21 days, followed by surgery.
  Interventions: Drug: docetaxel, cisplatin, 5 fluorouracil

INTERVENTIONS:
Drug: docetaxel, cisplatin, 5 fluorouracil
  Other Names: taxotere, cisplatin, tolerak

SUMMARY:
This is a phase II study of preoperative chemotherapy with docetaxel, cisplatin and 5-fluorouracil (TPF) in locally advanced resectable oral cavity squamous cell cancer. The aim is to improve the rate of pathological complete response to induction chemotherapy in a molecular enriched population, consisting of patients with tumour harbouring a functional p53 protein and/or showing low expression of beta-tubulin II.

DETAILED DESCRIPTION:
Patients with stage T2 (> 3 cm) T3 N1-N3 and T4a any N primary OCSCC are considered for enrolment in this trial. Patients will be asked to sign the informed consent for being admitted to the clinical study and in order to analyze the tumour biopsy. If a functional p53 protein status and/or low expression of beta-tubulin II is identified, patient will be enrolled in therapeutic part of the study. In case of different molecular profile, patient will not be enrolled in the study. A radiological work up of disease is required before to start CT. A magnetic resonance imaging (MRI) with DWI, and if available, a dynamic contrast enhanced (DCE)-MRI will be performed before therapy.

Each patient will receive induction CT, consisting of TPF (docetaxel 75 mg/sm and cisplatin 80 mg/sm day 1 and 5 fluorouracil 800 mg/sm each day in continuous infusion day 1-4, according to Paccagnella et al, ASCO 2008) for 3 cycles every 21 days, followed by surgery. Prophylactic antibiotic with ciprofloxacin 500 mg 2 times/day will be administered starting from day 5th to day 15th after each cycle; G-CSF is admitted as secondary prophylaxis in case of febrile neutropenia or neutropenia grade 4 at previous cycle. Patient will have clinical examination at baseline and before each CT cycle. Whenever a clinical suspicion of progressing disease will exist, a radiological restaging with MRI will be performed and in case of radiological progression according to RECIST 1.1 the patient will be submitted to surgical excision of the tumour. However, in any case the investigators may 14 judge that the disease is progressing and they consider that chemotherapy is no more indicated, the patient will be submitted to surgery even without a radiological confirmation of progression. In case of clinical SD or PR, a radiological restaging will be planned with MRI and DWI-MRI at least two weeks after the third cycle (a DWI- MRI and, if available a DCE-MRI, will be performed after 1st cycle in order to evaluate early response imaging). Surgery will be performed within one month after the last cycle of CT, if there are no clinical contraindications. After the surgical treatment, adjuvant treatment will be delivered according to recognized pathological risk factors (Bernier J, 2005). Patients will be followed up according to the Institutional follow-up policy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Males and females age > 18 years
* Histologically proved primary oral cavity squamous cell cancer (tumour extending to oropharynx are accepted if oropharyngeal invasion is < 20% of the tumour size)
* Stage T2 (T2 stage is accepted if tumour size is 3 cm or larger).-T3, N1- N3 and T4a any N
* WHO performance status < 1
* Availability of block of Formalin Fixed Paraffin Embedded (FFPE) biopsy of the tumour
* Radiological imaging of the tumour with MRI pre-therapy
* Effective contraception for both male and female subjects if risk of conception exists

Exclusion Criteria:

* Prior antitumour therapy for head & neck cancer (chemotherapy or biological therapy and radiotherapy)
* Metastatic disease
* Medical condition that contraindicate administration of TPF scheme, in particular:

  1. clinically significant cardiac disease including unstable angina, acute myocardial infarction in the previous 2 years, congestive heart failure and arrhythmia requiring therapy
  2. chronic or current infectious disease that contraindicate administration of chemotherapy causing neutropenia; known HIV, Hepatitis B or C positivity
  3. uncontrolled renal, hepatic, neurological, cerebral, psychiatric, haematological, gastrointestinal, pulmonary, vascular or endocrine diseases that could interfere with antiblastic treatment
* Pre-existing peripheral neuropathy according to Common Toxicity Criteria (CTC) Adverse Event grade > 1
* Pre-existing ototoxicity grade > 1
* Previous diagnosis of other cancer in the last 3 years (in situ cervical cancer or completely excised basocellular/squamocellular skin cancer are always admitted )
* Previous other cancer in oral cavity to less than 2 cm from existing primary
* Breast feeding women or women with a positive pregnancy test at Visit 0 or 1
* Screening laboratory values:

  * Neutrophils < 1.5 x 109/L
  * Platelets < 100 x 109/L
  * ALT or AST > 2.5 times upper limit of normal
  * Calculated creatinine clearance < 60 mL/min
  * Weight loss more than 20% in 3 months preceding the study
  * Technical unresectability defined as: T4b staging or N ulcerating the skin or encasing internal carotid

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-06; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
pathologic complete remission | After 9 weeks since chemotherapy start
  For what concerns primary endpoint of pathologic complete remission achievement, the patients will be assessed at time of surgery, i.e., after about 9 weeks since chemotherapy start.

SECONDARY OUTCOMES:
Progression free survival | 5 years
  Patients will be followed up to 5 years for what concerns PFS
Overall Survival | 5 years
  Patients will be followed up to 5 years for what concerns OS
Compliance to induction chemotherapy | 9 weeks
  Evaluation in terms of the number of cycles administered, actual and total doses dministered, dose modifications, delays and omissions, as well as reasons for deviation from planned therapy and overall treatment duration will be described
Percentage of patient receiving postoperative radiotherapy and chemotherapy | 6 months
  Patients will be followed for what concerns PFS, defined as the time from the date of randomization up to the date of first progression, second primary malignancy or death from any cause, whichever comes first.
Early functional response evaluation by DWI and DCE MRI | 3 weeks
  radiological evaluation after 1 cycle of induction chemotherapy
Comparison between (DWI - DCE) MRI response and pathological response | 9 weeks
  comparison between radiological assessment of response and pathological one

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Licitra, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori - Milan
Locations (1):
- Istituto Nazionale Tumori, Milan, Italy